CLINICAL TRIAL: NCT06994182
Title: Perspectives of Italian Employers Regarding the Return to Work Process of Employees Who Received a Cancer Diagnosis: a Qualitative Study
Acronym: employers_2024
Status: Recruiting | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Collaborators: Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC) (Other)
Responsible Party: Sponsor
Other Study IDs: 632/2024/OSS/AUSLRE
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Cancer Survivors
Keywords: Cancer Survivors; Return to work; Employers; Qualitative Research

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Employers: This cohort includes employers of active companies located in the province of Reggio Emilia. The Chamber of Commerce dell 'Emilia will provide a random list of the active company based on the type of company (profit, non-for-profit), type of sector (i.e., manufacturing, constructions), and number of employees (small, medium, large) to guarantee the representativeness of our context.

SUMMARY:
European Cancer Mission calls attention to the return to work (RTW) of cancer survivors (CSs), as one of the pivotal issues of the cancer continuum that need to be addressed through proper and prompt actions and recommendations. Employers are important stakeholders, as they can provide emotional and practical support, sustain communication during the entire process, and guarantee a gradual work reintegration. In Italy there is lack of knowledge regarding this topic. Thus, further exploration of Italian employers' perspectives on the RTW of employees with cancer should be performed to comprehend their unknown experiences.

The aim is to explore the perspectives of employers who dealt with the RTW process of employees who received a cancer diagnosis through a qualitative research design.

DETAILED DESCRIPTION:
Data collection will be performed through individual semi-structured interviews. Each interview will last around 60 minutes, and it can be arranged in person or remotely, depending on the participant's preference. Socio-demographic data, expertise of the employer, and company-related data will be collected through a semi-structured interview.

Experiences of employers will be collected through open-ended questions using an interview guide that was written based on the one used by Tiedtke et al., 2017, by adding some questions related to the facilitators and barriers perceived by employers during the sickness absence and RTW of employee with cancer.

The open-ended questions will concern general information about the company, employers' experience after cancer disclosure and during sick leave, employers' experience to sustain the RTW process and the long-term work reintegration, and the influence of the experience on the company.

Each interview will be audio-recorded, transcribed verbatim and analyzed according to the thematic analysis method using an inductive approach with open coding.

Analysis will be iterative and involve multiple researchers to ensure inter-rater reliability of the coding procedure and the methodological rigor of the analysis.

Themes generated will be discussed with Dutch researchers from the Amsterdam University Medical Centers.

Analyses will be carried out at the end of each interview because, based on the themes that will emerge from each interview, we will understand when to stop recruiting.

ELIGIBILITY:
Inclusion Criteria:

1. employers* of a company
2. being directly involved in managing the RTW process of at least one employee with cancer diagnosis in the last 5 years.

   * An employer can be the specific person who represents the company where the employee was working at the time of cancer diagnosis or a person who supported the employee during the sickness absence and the RTW process (e.g., line manager, human resource manager).

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of employers of the province of Reggio Emilia who managed the RTW process of employees with a cancer diagnosis. This population includes employers from companies with diverse characteristics (type of company and sector, and number of employees) to collect the perspectives of employers working in different settings.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
1. Open-ended questions of a semi-structured interview to collect the employers experience of the management of the RTW process | 12 months
  Themes describing how employers managed the RTW process of employees with cancer, of their feeling and thoughts, of what actions did they do, and of the relationships and communication with the other members of the company
Open-ended questions of a semi-structured interview to collect the employers' necessities while supporting the RTW process | 12 months
  Themes describing what employers require to support employees who receive a cancer diagnosis in the RTW process
Open-ended questions of a semi-structured interview to collect the employers perceived barriers and facilitators while supporting the RTW process | 12 months
  Themes describing the facilitators and barriers perceived by employers during the RTW process of employees who received a cancer diagnosis. For this outcome, themes will be classified using the Resource Dependence Institutional Cooperation (RDIC) model, developed by Rijk et al. and adjusted by Greidanus et al. (2018).

CONTACTS AND LOCATIONS:
Overall Officials: Sara Paltrinieri, PhD, OT, Principal Investigator — Azienda USL - IRCCS di Reggio Emilia
Locations (1):
- Azienda USL IRCCS di Reggio Emilia, Reggio Emilia, RE, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greidanus MA, de Boer AGEM, de Rijk AE, Tiedtke CM, Dierckx de Casterle B, Frings-Dresen MHW, Tamminga SJ. Perceived employer-related barriers and facilitators for work participation of cancer survivors: A systematic review of employers' and survivors' perspectives. Psychooncology. 2018 Mar;27(3):725-733. doi: 10.1002/pon.4514. Epub 2017 Sep 6. PMID 28753741
- [Background] Lawler M, De Lorenzo F, Lagergren P, Mennini FS, Narbutas S, Scocca G, Meunier F; European Academy of Cancer Sciences. Challenges and solutions to embed cancer survivorship research and innovation within the EU Cancer Mission. Mol Oncol. 2021 Jul;15(7):1750-1758. doi: 10.1002/1878-0261.13022. Epub 2021 Jun 15. PMID 34053182
- [Background] Paltrinieri S, Fugazzaro S, Bertozzi L, Bassi MC, Pellegrini M, Vicentini M, Mazzini E, Costi S. Return to work in European Cancer survivors: a systematic review. Support Care Cancer. 2018 Sep;26(9):2983-2994. doi: 10.1007/s00520-018-4270-6. Epub 2018 May 29. PMID 29845421
- [Background] de Rijk A, Amir Z, Cohen M, Furlan T, Godderis L, Knezevic B, Miglioretti M, Munir F, Popa AE, Sedlakova M, Torp S, Yagil D, Tamminga S, de Boer A. The challenge of return to work in workers with cancer: employer priorities despite variation in social policies related to work and health. J Cancer Surviv. 2020 Apr;14(2):188-199. doi: 10.1007/s11764-019-00829-y. Epub 2019 Nov 22. PMID 31758518
- [Background] Tiedtke CM, Dierckx de Casterle B, Frings-Dresen MHW, De Boer AGEM, Greidanus MA, Tamminga SJ, De Rijk AE. Employers' experience of employees with cancer: trajectories of complex communication. J Cancer Surviv. 2017 Oct;11(5):562-577. doi: 10.1007/s11764-017-0626-z. Epub 2017 Jul 14. PMID 28710544